CLINICAL TRIAL: NCT00583882
Title: A Prospective, Randomized Study to Evaluate the Risks Related to Central Venous Catheter Replacement Strategies in Patients With Acute Burn Injury
Brief Title: Central Venous Catheter Replacement Strategies in Patients With Acute Burn Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Michael S. O'Mara, Shriners Hosptial for Children Northern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200614292-1
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2008-01-02 (Estimated); Status verified 2007-12

CONDITIONS: Burns
Keywords: Central Venous Catheter; Guidewire; Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Change every 6 days, rewire every 6 days
  Interventions: Other: Routine change of central venous catheters
- 2 (Other): New site every 6 days
  Interventions: Other: Routine change of central venous catheters
- 3 (Other): New site every 12 days
  Interventions: Other: Routine change of central venous catheters

INTERVENTIONS:
Other: Routine change of central venous catheters — Changeing CVCs on a regular basis to decrease infection rate.

SUMMARY:
This project proposes to answer the following questions:

To determine the incidence of infection with three primary schedules of central venous catheter exchange in pediatric burn patients and to determine the regimen that will minimize infectious risk in children with burns.

The scientific knowledge to be acquired through this project is of likely benefit to the care of children with orthopaedic problems, spinal cord injuries or burns as follows:

The intention is to improve the outcomes in burned children by minimizing one of the most frequent causes of infection in the burn intensive care unit, those from central venous catheters. Decreasing infections will decrease morbidity, decrease length of stay, decrease costs, and decrease mortality in burned children

DETAILED DESCRIPTION:
Aim: To determine the incidence of infection with three primary schedules of central venous catheter exchange in pediatric burn patients and to create a system that will minimize infectious risk in this patient population.

Hypothesis: A strategy of routine catheter changes without guidewire exchange will result in no more infections and a decreased risk of mechanical complications over frequent guidewire exchange or frequent new-site replacement.

Background: Reviews of burned children have implied that it is safe to change CVCs on a weekly basis, either by new site insertion or by wire exchange. In non-burn populations the routine use of wire exchange may increase infectious risk. Laboratory investigations have shown that the longer catheters are in place, the more often they are colonized with bacteria; this translates to an increase in catheter infection and patient sepsis. Centers for Disease Control recommendations note that catheters should not be routinely changed. The burn literature has disagreed with this concept, proffering that the change in microbial milieu from the burn wound increases infection risk, and national data indicates that burn units have three to four times higher rates of catheter related bloodstream infections than do other intensive care units. There is a trend in the existent retrospective data that using wires to change central venous catheters increases the risk of infection: CVCs changed to a new site have an infection rate of 16.6 per 1000 catheter days, whereas those changed by means of a wire have a rate of 25.2 per 1000 catheter days.

Methods: Patients will be randomized to three intervention groups: a frequent (6 days) moving of catheters to new sites; an alternating schedule of wire exchanges and new sites (every 6 and 12 days); and a less frequent moving of catheters to new sites (12 days) without wire exchange. This project requires enough patients to show a difference between three intervention groups. A significant decrease in infection rate would be from the current 20 infections per 1000 catheter days to approximately 15 per 1000 catheter days. This would require a minimum of 1000 catheter days per group.

ELIGIBILITY:
Inclusion Criteria:

* Burn patient with central venous catheter

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
CVC related blood stream infections. | patient discharge/CVC removal

SECONDARY OUTCOMES:
CVC mechanical complications | patient discharge/CVC removal

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospital for Children Northern California, Sacramento, California, United States